CLINICAL TRIAL: NCT01106807
Title: Exploratory Study to Evaluate the Efficacy and Safety of CD07223 1.5% Gel and 0.5% Gel in Subjects With Acne
Brief Title: Exploratory Study to Evaluate the Efficacy and Safety of CD07223 Gel in Subjects With Acne
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD.06.SPR.18173
Record Dates: First submitted 2010-04-19; First posted 2010-04-20 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2012-04

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination; Adapalene; Benzoyl Peroxide; Gels

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- CD07223 1.5% gel (Experimental): 500 microliters of CD07223 1.5% gel on one half-face twice daily for six weeks and Epiduo vehicle gel on the other half-face
  Interventions: Drug: Epiduo vehicle gel; Drug: CD07223
- CD07223 0.5% gel (Experimental): 500 microliters of CD07223 0.5% gel on one half-face twice daily for six weeks and Epiduo vehicle gel on the other half-face
  Interventions: Drug: Epiduo vehicle gel; Drug: CD07223
- Epiduo (adapalene and benzoyl peroxide) 0.1%/2.5% gel (Active Comparator): 500 microliters of Epiduo (adapalene and benzoyl peroxide) 0.1%/2.5% gel on one half-face and 500 microliters of the Epiduo vehicle gel on the other half-face in the morning and in the afternoon, 500 microliters of Epiduo vehicle gel on both half-faces
  Interventions: Drug: Epiduo vehicle gel; Drug: Epiduo (adapalene and benzoyl peroxide) 0.1%/2.5% gel

INTERVENTIONS:
Drug: Epiduo vehicle gel — 500 microliters of Epiduo vehicle gel on one half-face twice daily for six weeks
Drug: CD07223 — 500 microliters of CD07223 1.5% gel on one half-face twice daily for six weeks
  Arms: CD07223 1.5% gel
Drug: CD07223 — 500 microliters of CD07223 0.5% gel on one half-face twice daily for six weeks
  Arms: CD07223 0.5% gel
Drug: Epiduo (adapalene and benzoyl peroxide) 0.1%/2.5% gel — 500 microliters Epiduo Gel on one of the half-face for the morning dose
  Arms: Epiduo (adapalene and benzoyl peroxide) 0.1%/2.5% gel

SUMMARY:
The purpose of the study is to evaluate the efficacy of CD07223 1.5% Gel and 0.5% gel in reducing inflammatory, non-inflammatory, and total acne lesion counts after 6 weeks of twice daily applications. The study will also evaluate the safety of the study products using tolerance and adverse event data.

ELIGIBILITY:
Inclusion Criteria:

* subject has a clinical diagnosis of acne vulgaris with facial involvement
* the subject has at least 15 inflammatory lesions and 25 non-inflammatory lesions (excluding the nose) but no more than 2 nodules on the face

Exclusion Criteria:

* subject has a severe acne form or secondary acne form
* the number of inflammatory or non-inflammatory lesions on one half-face is greater than twice the number on the other half-face
* the subject has a known allergy or sensitivity to any of the components of the study products
* subject is not willing to respect wash-out periods for topical and/or systemic treatments

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Total acne lesion count | 6 weeks
  change in total number of acne lesion count from baseline to end of treatment
Percent change of acne lesion count | 6 weeks
  Percent change of acne lesion count from baseline to end of treatment

SECONDARY OUTCOMES:
Lesion counts- Inflammatory | 6 weeks
  change in lesion count from baseline at each evaluation visit; efficacy preference at the end of treatment by investigator and subject
Lesion count- non-inflammatory | 6 weeks
  change in lesion count from baseline at each evaluation visit; efficacy preference at the end of treatment by investigator and subject
Lesion counts- Inflammatory | 6 weeks
  Percent change of acne lesion count from baseline at each evaluation visit
Lesion count- non-inflammatory | 6 weeks
  Percent change of acne lesion count from baseline at each evaluation visit

CONTACTS AND LOCATIONS:
Overall Officials: Michael Graeber, MD, Study Director — Galderma R&D
Locations (9):
- United States (9):
  - Burke Pharmaceuticals, Hot Springs, Arkansas
  - Dermatology Specialist PSC, Louisville, Kentucky
  - Grekin Skin Institute, Warren, Michigan
  - TKL Research, Rochelle Park, New Jersey
  - Piedmont Medical Research, Winston-Salem, North Carolina
  - Cetero, Fargo, North Dakota
  - Derm Research, Inc, Austin, Texas
  - J & S Studies, Bryan, Texas
  - Education and Research Foundation, Inc, Lynchburg, Virginia